CLINICAL TRIAL: NCT07035379
Title: A Phase I/II Study Evaluating the Safety, Tolerability, Pharmacokinetics and Anti-Tumor Activity of TRS005 in Combination With Cyclophosphamide, Doxorubicin, and Prednisone（T-CHP） in Previously Untreated Patients With CD20-positive DLBCL
Brief Title: A Phase I/II Study of TRS005 in Combination With Cyclophosphamide, Doxorubicin, and Prednisone（T-CHP） in Previously Untreated Patients With CD20-positive DLBCL
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhejiang Teruisi Pharmaceutical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRS00501003
Record Dates: First submitted 2025-06-13; First posted 2025-06-25 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-06

CONDITIONS: Diffuse Large B-Cell Lymphoma (DLBCL)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Cyclophosphamide; Doxorubicin; Prednisolone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TRS005+CHP (Experimental): TRS005 in Combination With Cyclophosphamide, Doxorubicin, and Prednisone（T-CHP）
  Interventions: Drug: TRS005; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisolone

INTERVENTIONS:
Drug: TRS005 — TRS005 will be administered at a starting dose of 0.8mg/kg IV every 3 weeks (starting from Cycle 1 Day 1), for 6 cycles (up to 8).
Drug: Cyclophosphamide — Cyclophosphamide will be administered at 750 milligrams per square meter (mg/m^2) IV every 3 weeks (starting from Cycle 1 Day 1), for 6 cycles.
Drug: Doxorubicin — Doxorubicin will be administered at 50 mg/m^2 IV every 3 weeks (starting from Cycle 1 Day 1), for 6 cycles.
Drug: Prednisolone — Prednisolone will be administered at 100 mg orally daily for 5 days every 3 weeks (starting from Cycle 1 Day 1), for 6 cycles.

SUMMARY:
This trial is a multicenter, open-label, single-arm, dose-escalation and dose-expansion clinical trial. The dose was increased according to the "3 + 3" rule. Patients with previously untreated patients with CD20-positive DLBCL were selected to evaluate the safety, tolerance (DLT, MTD), pharmacokinetics, and anti-tumor activity of TRS005 in combination with standard doses of cyclophosphamide, doxorubicin, and prednisone（T-CHP） by intravenous drip every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 1. Part I: Age 18 -65 years old; Part II: Aged ≥ 18 years old, both male and female.
* 2. Previously untreated patients with CD20-positive DLBCL diagnoses by 2022 WHO.
* 3. Measurable disease of at least 15mm (node)/10mm (extranodal).
* 4. ECOG performance status 0-2.
* 5. International Prognostic Index (IPI) score of 2-5.
* 6. Estimated survival time ≥6 months.
* 7. Having sufficient organ function.
* 8. Female and male patients of childbearing age and their spouses are willing to carry out adequate contraception throughout the study period, and female patients of childbearing age must have negative serum pregnancy test within 7 days before the first administration.
* 9. Patients voluntarily agree to participate in the study and to sign the informed consent form.

Exclusion Criteria:

* 1. Contraindication to any of the individual components of study drugs, including prior receipt of xenoproteins, biological agents.
* 2. Serologic evidence of chronic hepatitis B virus (HBV) infection and unable or unwilling to receive standard prophylactic antiviral therapy or with detectable HBV viral load; Serologic evidence of hepatitis C virus (HCV) infection without completion of curative treatment or with detectable HCV viral load; Human immunodeficiency virus (HIV) seropositive.
* 3. Clinically apparent central nervous system (CNS) lymphoma.
* 4. Patient has ≥ Grade 2 peripheral neuropathy.
* 5. Investigator-assessed diabetes uncontrolled by drug therapy.
* 6. Clinically significant third space fluid accumulation.
* 7. Patients with other malignancies within the past 5 years.
* 8. With active autoimmune diseases.
* 9. Accompanied by serious cardiovascular diseases.
* 10. Accompanied by serious diseases and serious active infections.
* 11. The dosage of steroid hormone (prednisone phase equivalent) used greater than 20mg/ day within 28 days prior to first administration for more than 14 consecutive days, or immunosuppressive treatment.
* 12. Various vaccines were inoculated within 28 days prior to first administration;
* 13. Major surgery (except diagnostic biopsy) within 28 days prior to first administration or during the study period.
* 14. Participate in clinical trials of other drugs or medical devices within 28 days prior to first administration.
* 15. Serious medical or psychiatric illness likely to interfere with participation in this study.
* 16. Investigators assessed as unsuitable to participate in this study for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Part I: Dose Limiting Toxicities (DLTs) and Maximum Tolerated Dose (MTD) | Cycle 1 Day 1 (C1D1) to Cycle 1 Day 21 (C1D21)
  All dose-escalation cohorts will consist of at least 3 participants. If a DLT is observed in 1 participant at a given dose level during the DLT observation period before dose escalation, additional participants will be enrolled at that dose level for a total of at least 6 participants. DLT assessment forms part of determining the Maximum Tolerated Dose (MTD). The highest dose level resulting in DLTs in less than one-third of a minimum of 6 participants will be declared the MTD.
Part I and II: Adverse Events | Day 1 up to approximately 6 months
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events. AEs were reported based on the national cancer institute common terminology criteria for AEs, Version 5.0 (NCI-CTCAE, v5.0). Reported are the number of subjects with AEs, Grade 3-5 AEs, and Serious Adverse Events (SAEs).

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | At the end of treatment (Month 6)
  The overall response rate (ORR) was defined as the proportion of participants achieving complete response (CR) or partial response (PR) based on Lugano 2014 criteria
Duration of Response (DOR) | Up to 24 months
  Duration of Overall Response (DOR), estimated using the Kaplan Meier method, is measured from Lugano 2014 criteria are met for CR or PR (whichever is first recorded) , until the first date that recurrent or progressive disease is objectively documented. Patients without progressive disease are censored at the date of last disease assessment.
Progression-Free Survival (PFS) | Up to 24 months
  Progression-free survival based on the Kaplan-Meier method is defined as the duration between randomization and documented disease progression (PD) per Lugano criteria or death, or is censored at time of last disease assessment.
Overall Survival (OS) | Up to 24 months
  Overall Survival (OS) based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Immunogenicity | At the end of treatment (Month 6)
  ADA will be assessed in all participants. NAb will be assessed in samples that are ADA positive.
Serum concentration | At the end of cycle 4 (each cycle is 21 days)
  Total TRS005, TRS005 unconjugated MMAE, and antibody-conjugated Mono-Methyl Auristatin E [acMMAE]

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences, Cancer Hospital, Beijing, Beijing Municipality, China